CLINICAL TRIAL: NCT01180478
Title: A Multi-center, International Study to Compare Use of Narrow Band Imaging (NBI) Versus White Light(WL) During Transurethral Resection of Bladder Tumors (TURB) to Asses Recurrence of Bladder Cancer in Terms of Safety and Efficacy
Brief Title: Comparison Study of Narrow Band Imaging Versus White Light Resection in Patients With Bladder Tumors/Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Office of the Endourological Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-004660
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Results first posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Urothelial carcinoma; Stage pTa or pT1; NMIBC Ta/T1; Narrow Band Imaging; White Light Cystoscopy; Transurethral resection; Superficial bladder tumor; Positive urine cytology
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrow Band Imaging (Other): Narrow Band Imaging (NBI)
  Interventions: Device: Narrow Band Imaging
- White Light Trans Urethral Resection (Other): White Light Trans Urethral Resection
  Interventions: Device: White Light

INTERVENTIONS:
Device: White Light — White Light Cystoscopy
  Arms: White Light Trans Urethral Resection
Device: Narrow Band Imaging — Narrow Band Imaging
  Arms: Narrow Band Imaging

SUMMARY:
The purpose of this study is to compare the recurrence rate at 1 year following Narrow Band Imaging and trans-urethral resection of bladder tumor with White Light and TURB in patients with non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
Currently bladder tumors are diagnosed visually with standard cystoscopy that uses white light, or light that is generated encompassing the entire visual spectrum. Some tumors such as carcinoma in situ may not be visible using white light and require patients to undergo random bladder biopsies in order to find the cancer. Recently the development of photodynamic agents have been shown to enhance these procedures to accomplish better resection and identify over-looked tumors. However, these methods often require the instillation of dyes into the bladder as well as specialized cystoscopes. Narrow band imaging (NBI) is now available which uses a special filter to limit the light to only certain wavelengths which allows the identification of areas of increased vascularity or abnormalities without the need for dyes. NBI has been investigated in gastro-intestinal disease and found to be beneficial. Early reports in urology suggest that this technology may reduce the number of tumors that are missed which could impact the recurrence rate of bladder tumors, but this is not known at this time.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for treatment of primary or recurrent non-muscle invasive bladder cancer
* Patients greater than 18 years of age
* No tumors in the upper tract (kidneys or ureters)
* No previous pelvic radiation

Exclusion Criteria:

* Gross hematuria at the time of resection making visualization with NBI not possible
* Participation in other clinical studies with investigations drugs concurrently or within 30 days.
* Pregnancy
* Conditions associated with a risk of poor compliance or unwilling to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 965 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean de la Rosette, MD, Study Director — AMC University Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Narrow Band Imaging | White Light Trans Urethral Resection
Started | 484 | 481
Completed | 303 | 293
Not Completed | 181 | 188

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrow Band Imaging | White Light Trans Urethral Resection | Total
Number analyzed (Participants) | 484 | 481 | 965
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (12.5) | 66.7 (12.3) | 66.24 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 98 | 192
  Male | 390 | 383 | 773
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 4 | 8 | 12
  Canada | 52 | 40 | 92
  China | 41 | 34 | 75
  Czechia | 51 | 67 | 118
  Hong Kong | 23 | 17 | 40
  India | 14 | 13 | 27
  Italy | 3 | 10 | 13
  Japan | 97 | 75 | 172
  South Korea | 43 | 48 | 91
  Norway | 13 | 16 | 29
  Romania | 29 | 30 | 59
  Russia | 9 | 13 | 22
  Spain | 9 | 13 | 22
  Netherlands | 41 | 38 | 79
  Turkey | 38 | 39 | 77
  United States | 11 | 17 | 28
  United Arab Emirates | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence and Recurrence Rate at 1 Year Following Narrow Band Imaging and TURB (Arm A) Versus White Light Trans Urethral Resection of Bladder Cancer (TURB) (Arm B) in Patients With Non Muscle Invasive (pTa/T1) Bladder Cancer.
Description: The primary outcome measure was recurrence rate at 1 year. A recurrence was defined as the new occurrence of a bladder cancer at the same site as or at a different site from the index cancer.
Time Frame: 1 year after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging | White Light
Number analyzed (Participants) | 484 | 481
Participants | 104 | 109
Statistical Analysis 1: Comparison: Narrow Band Imaging vs White Light; The expected recurrence rate in the WL-assisted TURBT group was 35%.14 To detect a clinically relevant difference in recurrence detection rates ≥10% at a 5% significance level and a power of 80%, the required sample size per treatment was calculated to be 329 patients (658 patients in total); Test type: Superiority or Other; p = 0.585, Log Rank

2. Secondary Outcome: Number of Participants With Persistence/Recurrence of Tumors at First 3 Month Follow up After NBI Versus WL Cystoscopy and Tumor Resection
Time Frame: 3 months after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging | White Light Trans Urethral Resection
Number analyzed (Participants) | 484 | 481
Participants | 59 | 61
Statistical Analysis 1: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Test type: Superiority or Other; p = 0.742, Chi-squared

3. Secondary Outcome: Peri-operative Morbidity (30 Days) of TURB Between NBI and WL Resection Using the Clavien System.
Description: Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.
  Grade II Requiring pharmacological treatment with drugs other than those allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III Requiring surgical, endoscopic or radiological intervention Grade III-a Intervention not under general anaesthesia Grade III-b Intervention under general anaesthesia
  Grade IV Life-threatening complication (including CNS complications: brain haemorrhage, ischaemic stroke, subarachnoid bleeding, but excluding transient ischaemic attacks) requiring IC/ICU management Grade IV-a Single organ dysfunction (including dialysis) Grade IV-b Multi-organ dysfunction
  Grade V Death of a patient
Time Frame: 30 days
Population: The Clavien grading of perioperative complications variable contains missings, therefore the valid percentages are presented in the outcome measure data table. The NBI group had 2 missing values, and the WL group had 3 missing values. Therfore, the overall number deviates from 484 and 481.
  Below shown is a categorical variable with 8 categories
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging | White Light Trans Urethral Resection
Number analyzed (Participants) | 482 | 478
Participants
  None | 415 | 429
  I | 28 | 19
  II | 23 | 21
  IIIA | 11 | 4
  IIIB | 3 | 5
  IVA | 0 | 0
  IVB | 0 | 0
  V | 2 | 0
Statistical Analysis 1: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; The statistical analyses refers to comparison of the different 8 categories (one variable) mentioned of the Clavien grading of perioperative complications between Narrow Band Imaging and White Light Trans Urethral Resection; Test type: Superiority or Other; p = 0.170, Fisher Exact; The analysis was performed by using the Fisher exact test, because the criteria for using the Chi square test were not met

4. Secondary Outcome: Risk Factors for the Development of Peri-operative Morbidity After Instrumental Treatment.
Description: We looked at different perioperative complications in order to discover peri-operative morbidity after instrumental treatment. The following variables were analyzed: Bleeding, Fever, UTI, Bladder cramps, DVT, CVA/TIA, Lung embolism, Sepsis, Acute Abdomen, and Other perioperative complications.
Time Frame: peri-operative
Population: The variables contain missing values, therefore the numbers in the below table differs from the overall numbers reported
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging | White Light Trans Urethral Resection
Number analyzed (Participants) | 484 | 481
Participants
  Bleeding: number analyzed (Participants) | 431 | 414
  Bleeding | 36 | 27
  Fever: number analyzed (Participants) | 422 | 407
  Fever | 9 | 7
  UTI: number analyzed (Participants) | 422 | 404
  UTI | 8 | 10
  Bladder cramps: number analyzed (Participants) | 423 | 407
  Bladder cramps | 19 | 10
  DVT: number analyzed (Participants) | 421 | 404
  DVT | 0 | 0
  CVA/TIA: number analyzed (Participants) | 420 | 404
  CVA/TIA | 2 | 0
  Lung embolism: number analyzed (Participants) | 421 | 404
  Lung embolism | 0 | 0
  Sepsis: number analyzed (Participants) | 421 | 404
  Sepsis | 2 | 0
  Acute Abdomen: number analyzed (Participants) | 421 | 403
  Acute Abdomen | 1 | 1
  Other perioperative complication: number analyzed (Participants) | 421 | 406
  Other perioperative complication | 9 | 13
Statistical Analysis 1: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison of the numbers in 'Bleeding' between NBI and WL; Test type: Superiority or Other; p = 0.311, Chi-squared
Statistical Analysis 2: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison of the numbers in 'Fever' between NBI and WL; Test type: Superiority or Other; p = 0.666, Chi-squared
Statistical Analysis 3: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'UTI' between NBI and WL; Test type: Superiority or Other; p = 0.569, Chi-squared
Statistical Analysis 4: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'Bladder cramps' between NBI and WL; Test type: Superiority or Other; p = 0.111, Chi-squared
Statistical Analysis 5: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'DVT' between NBI and WL; Test type: Superiority or Other; Non of the participants/patients had DVT. Therefore, the p-value is not available
Statistical Analysis 6: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'CVA/TIA' between NBI and WL; Test type: Superiority or Other; p = 0.500, Fisher Exact
Statistical Analysis 7: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'Lung embolism' between NBI and WL; Test type: Superiority or Other; Non of the participants/patients had a lung embolism. Therefore, no p-value was available
Statistical Analysis 8: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'Sepsis' between NBI and WL; Test type: Superiority or Other; p = 0.500, Fisher Exact
Statistical Analysis 9: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'Acute Abdomen' between NBI and WL; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 10: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Comparison in the number of 'Other perioperative complication' between NBI and WL; Test type: Superiority or Other; p = 0.170, Chi-squared

5. Secondary Outcome: Recurrence Rate Related to Additional Treatment Following TURB.
Time Frame: Until 135 days
Population: Only 61 of the patients in the total population in the NBI group, and 69 of the patients in the total population of the WL group received a Re-TURBT after initial TURBT (within 135 days). These numbers therefore differ and deviate from the Participant Flow module.
Measure: Number; unit: participants
Arm/Group | Narrow Band Imaging | White Light Trans Urethral Resection
Number analyzed (Participants) | 61 | 70
participants | 27 | 27
Statistical Analysis 1: Comparison: Narrow Band Imaging vs White Light Trans Urethral Resection; Test type: Superiority or Other; p = 0.553, Chi-squared

ADVERSE EVENTS:
Description: Only Serious Adverse Events were monitored
Arm/Group | Narrow Band Imaging | White Light Trans Urethral Resection
Serious Adverse Events (participants affected / at risk) | 25/484 | 27/481
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Narrow Band Imaging (N=484) | White Light Trans Urethral Resection (N=481)
urinary tract infection (Infections and infestations) | 1 | 1
galbladder carcinoma (Hepatobiliary disorders) | 0 | 1
radical cystectomy (Renal and urinary disorders) | 1 | 0
lung adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hydronephrosis (Renal and urinary disorders) | 1 | 0
hip's fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
cardiogenic embolism (Vascular disorders) | 1 | 0
transurethral urethrotomy (Renal and urinary disorders) | 1 | 0
campylobacter colitis (Infections and infestations) | 0 | 1
rectorrhagia (Gastrointestinal disorders) | 0 | 1
patient died of intestinal obstruction (Gastrointestinal disorders) | 1 | 1
patient died of chest infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1
patient died of unknown cause (General disorders) | 2 | 2
cerebrovascular attack (Vascular disorders) | 1 | 0
patient died by car accident (Injury, poisoning and procedural complications) | 0 | 1
patient died of cardiac arrest (Cardiac disorders) | 1 | 1
patient died of bladder cancer (Renal and urinary disorders) | 2 | 5
obturator kick (Injury, poisoning and procedural complications) | 1 | 0
patient died by renal insuffiency and prostate cancer (Renal and urinary disorders) | 1 | 0
acute exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1
herniainguinalis (Gastrointestinal disorders) | 0 | 1
patient died of respiratory insuffiency by bilaterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pulmonary embolism (Vascular disorders) | 0 | 1
acute prostatitis (Infections and infestations) | 0 | 1
patient died of another neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
transurethral resection prostate (Renal and urinary disorders) | 0 | 1
transurethral urinary resection (Renal and urinary disorders) | 0 | 1
patient died of kidney failure (Renal and urinary disorders) | 0 | 1
patient died of heart attack (Cardiac disorders) | 1 | 0
urethral injury occurred at time of TUR (Injury, poisoning and procedural complications) | 1 | 0
patient died of cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
hematuria (Renal and urinary disorders) | 0 | 1
infection of unknown origin (Infections and infestations) | 0 | 1
euthanasia (General disorders) | 0 | 1
patient died of asystolia (Cardiac disorders) | 1 | 0
patient died of biliary tract cancer (Hepatobiliary disorders) | 1 | 0
patient died of pancreas cancer (Gastrointestinal disorders) | 1 | 0
patient died of septicaemia (Infections and infestations) | 1 | 0
radical cystectomy + bricker (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
There is a possibility of observer bias favouring NBI as a limitation of this single-blind study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No